CLINICAL TRIAL: NCT07106671
Title: A Prospective, Single-Arm, Single-Center, Phase II Clinical Trial of Siltuximab for Cytokine Release Syndrome and Immune Effector Cell-Associated Neurotoxicity After CAR-T Treatment in Multiple Myeloma
Brief Title: A Phase II Study of Siltuximab for CRS/ICANs After CAR-T in Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025006
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: CRS - Cytokine Release Syndrome; Myeloma
MeSH Terms: conditions — Cytokine Release Syndrome; Neoplasms, Plasma Cell | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Siltuximab (Experimental): Multiple myeloma patients with persistent grade 1 CRS/ICANS for 12 hours or grade ≥2 CRS/ICANS after CAR-T therapy will receive Siltuximab (11 mg/kg) immediately. If symptoms persist for another 12 hours, repeat Siltuximab and corticosteroids are allowed. If unresolved or worsened, rescue therapy with tocilizumab, corticosteroids, or other medications will be given.
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — Siltuximab 11mg/kg

SUMMARY:
This is a prospective Phase II study evaluating Siltuximab for CRS and ICANS after CAR-T infusion in multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be informed and voluntarily sign the Informed Consent Form (ICF).
2. Age ≥18 years old.
3. Diagnosed with multiple myeloma according to IMWG diagnostic criteria.
4. Developed CRS (grade ≥1) and/or ICANS (grade ≥1) after CAR-T treatment.

Exclusion Criteria:

1. Creatinine clearance <30 mL/min.
2. Platelet count <75,000/μL, absolute neutrophil count <1,000/μL, or hemoglobin <60 g/L at screening.
3. ALT or AST >3× ULN, or bilirubin >2× ULN.
4. Known severe cardiac conditions, including NYHA class III/IV heart failure, uncontrolled angina, arrhythmia, or hypertension, myocardial infarction within 6 months, or other uncontrolled/severe cardiovascular diseases, including prior cerebrovascular events with residual deficits.
5. Severe comorbidities, including active infections, known active HBV/HCV, HIV infection, uncontrolled diabetes, or serious conditions like chronic restrictive lung disease or cirrhosis.
6. Known intolerance to Siltuximab.
7. Known central nervous system (CNS) involement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete CRS resolution rate | 14 days
  14-day Complete CRS Resolution Rate: No CRS Symptoms for 24 Consecutive Hours

SECONDARY OUTCOMES:
CANS Resolution Rate | 28 day
  28-day ICANS Resolution Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China